CLINICAL TRIAL: NCT00849095
Title: As Needed Budesonide/Formoterol Combination Versus Regular Budesonide/Formoterol Combination Plus as Needed Terbutaline in Mild-Moderate Persistent Asthma
Brief Title: Prn Budesonide/Formoterol Versus Regular Budesonide/Formoterol Plus Prn Terbutaline in Mild-Moderate Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alberto Papi, MD, Professor, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIFA-ASMA-BF-001; EudraCT number: 2008-004127-36 (Registry Identifier: NCT00849095)
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Asthma
Keywords: Adult; Asthma; Bronchodilator Agents; Budesonide; Double-Blind Method; Drug Therapy, Combination; Ethanolamines; Female; Forced Expiratory Volume; Humans; Male; Terbutaline
MeSH Terms: conditions — Asthma | interventions — Budesonide; Terbutaline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- as needed medication (Experimental): patients assigned to this arm will take bid inhaled placebo plus prn inhaled 160/4.5 mcg budesonide/formoterol combination
  Interventions: Drug: budesonide/formoterol combination (PRN); Drug: placebo
- guideline treatment (Active Comparator): bid inhaled 160/4.5 mcg budesonide/formoterol combination plus prn 500 mcg terbutaline
  Interventions: Drug: budesonide/formoterol combination; Drug: terbutaline

INTERVENTIONS:
Drug: budesonide/formoterol combination (PRN) — budesonide/formoterol combination 160/4.5 mcg 1 inhalation used as needed for a period of 52 weeks
  Other Names: budesonide/formoterol combination
  Arms: as needed medication
Drug: budesonide/formoterol combination — budesonide/formoterol 160/4.5 mcg 1 inhalation bid
  Arms: guideline treatment
Drug: placebo — bid inhaled placebo
  Arms: as needed medication
Drug: terbutaline — as needed terbutaline 500 mcg for a period of 52 weeks
  Arms: guideline treatment

SUMMARY:
Study No.001 about Budesonide/Formoterol use in ASthMA sponsored by Agenzia Italiana del FArmaco (Italian Drug Agency) (AIFA-ASMA-BF-001) The aim of the study is to verify whether asthma not controlled by low doses inhaled corticosteroids, thus in need for step up therapy, can be equally controlled by guidelines recommended regular bid treatment with long acting beta agonist/inhaled corticosteroid (ICS/LABA) combination or the symptom driven use of an ICS/LABA combination in the absence of maintenance therapy. The study is designed to be able to evaluate the non inferiority of regular placebo plus prn inhaled budesonide/formoterol (experimental treatment) versus regular, twice daily 160/4.5 mcg inhaled budesonide/formoterol combination plus prn inhaled terbutaline (guidelines recommended treatment).

DETAILED DESCRIPTION:
Asthma is a problem worldwide, with an estimated 300 million affected individuals.There is evidence that asthma prevalence has been increasing in the last decades in some countries, including Italy. Analyses of the cost of asthma lead to conclude that the burden of the disease depend on the extent to which exacerbations are avoided since emergency treatment is more expensive than regular treatment.

Based on solid evidence, international guidelines recommend regular treatment with low dose ICS for mild persistent asthma and treatment with combination therapy [low dose ICS plus long-acting beta2-agonists (LABA)] for patients with asthma not controlled by low doses ICS alone. Recent studies have undermined the axiom that treatment with ICS must be regular to achieve and maintain asthma control, as equivalent control has been obtained either with prn use of an inhaled combination of a short acting beta2 agonist (SABA) and an ICS, or with a short course of 10 days high dose ICS at the start of exacerbations. In moderate-severe asthma regularly treated with inhaled ICS/LABA combination, the symptom-driven use of the same inhaled ICS/LABA combination as reliever is superior to the symptom-driven use of SABA or LABA alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female out-patient aged from 18 years to 65 years
* Clinical diagnosis of moderate persistent asthma for at least 6 months, according to GINA revised version 2006 guidelines
* Post-bronchodilator forced expiratory volume (FEV1) at least 80% of the predicted
* Either positive methacholine challenge test (PC20 FEV1< 4mg/ml or PD20 FEV1<0.8 mg) or positive response to the reversibility test in the last year
* Asthma either not adequately controlled with low-dose (≤500 mcg beclomethasone or equivalent) inhaled corticosteroids (ICS) or controlled by bid inhaled combination of low-dose ICS/long acting beta-2 agonists (LABA)
* A co-operative attitude and ability to be trained to correctly use the dry powder inhalator and to complete the diary cards
* Written informed consent obtained

Exclusion Criteria:

* Inability to carry out pulmonary function testing
* Moderate severe asthma associated with reduced lung function
* History of near-fatal asthma and/or admission intensive care unit because of asthma
* 3 or more courses of oral corticosteroids or hospitalization for asthma during the previous year
* Diagnosis of COPD as defined by the GOLD guidelines
* Evidence of severe asthma exacerbation or symptomatic infection of the airways in the previous 8 weeks
* Current smokers or recent (less than one year) ex-smokers, defined as smoking at least 10 pack/years
* History or current evidence of heart failure, coronary artery disease, myocardial infarction, severe hypertension, or cardiac arrhythmias
* Diabetes mellitis
* Percutaneous transluminal coronary angioplasty (PTCA) or coronary artery by-pass graft (CABG) during the previous six months
* Abnormal ECG
* Clinically significant or unstable concurrent diseases: uncontrolled hyperthyroidism, significant hepatic impairment, poorly controlled pulmonary disease (tuberculosis, active mycotic infection of the lung), gastrointestinal (e.g., active peptic ulcer), neurological or haematological autoimmune diseases
* Malignancy
* Any chronic diseases with prognosis < 2 years
* Pregnant or lactating females or not able to exclude pregnancy during the study period
* History of alcohol or drug abuse
* Patients treated with monoamine oxidase inhibitors, tricyclic antidepressants or beta-blockers as regular use
* Allergy, sensitivity or intolerance to study drugs and/or study drug formulation ingredients
* Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study
* Patients who received any investigational new drug within the last 12 weeks
* Patients who have been previously enrolled in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Actual)
Dates: Start 2009-04; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
comparison between groups of the relative risk for treatment failure | 52 weeks

SECONDARY OUTCOMES:
number of treatment failures | 52 weeks
time to first treatment failure | 52 weeks
differences between groups of lung function parameters, quality of life, symptoms score, use of as needed medication, adverse events | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Papi, MD, Principal Investigator — Università degli Studi di Ferrara
Locations (31):
- Italy (31):
  - Ospedale regionale Umberto I, Unità Operativa di Allergologia, Ancona, AN
  - Fondazione S. Maugeri - IRCCS -dipartimento di Pneumologia riabilitativa, Cassano delle Murge, BA
  - Dipartimento di Scienze Mediche-Unità Operativa di Pneumologia, Benevento, BN
  - Policlinico Sant'Orsola Malpighi, Unità Operativa di Pneumologia, Bologna, BO
  - Università degli Studi di Catania, Unità operativa di Pneumologia, Catania, CT
  - Università Magna Grecia Catanzaro, unità operativa di Pneumologia, Catanzaro, CZ
  - Ospedale Morgagni Pierantoni, azienda Ospedaliera di Forlì, Unitaà operativa di Pneumologia, Forlì, FC
  - UNIVERSITà DEGLI STUDI DI FERRARA, CLINICA DI MALATTIE DELL'APPARATO RESPIRATORIO, Ferrara, FE
  - Università degli studi di Foggia, ospedale pneumologico D'Avanzo, unità operativa di malattie dell'apparato respiratorio, Foggia, FG
  - Ospadale San Carlo Borromeo - Unità operativa di Pneumologia, Milan, MI
  - Ospedale città di Sesto San Giovanni, Unità operativa di Pneumologia, Sesto San Giovanni, MI
  - Università di Modena e Reggio Emilia, Unità operativa di Pneumologia, Modena, MO
  - Giuseppina Bertorelli, Parma, Parma
  - Università degli Studi di Palermo, Ospedale "V. Cervello", Palermo, Pa
  - Università degli studi di Padova, dipartimento di Pneunmologia, Padua, PD
  - Università degli studi di Padova, Medicina del Lavoro, Padua, PD
  - Università degli studi di Pisa, Ospedale Cisanello, unità operativa di Pneumologia, Pisa, PI
  - Università degli stiudi di Parma, unità operativa di Pneumologia, Parma, PR
  - IRCCS Fondazione S Maugeri, Dipartimento di Allergologia, Pavia, PV
  - Università degli studi di Pavia, dipartimento di Pneumologia, Pavia, PV
  - università Cattolica del Sacro Cuore, Columbus, unità operativa di allergologia, Roma, RM
  - Università Cattolica del Sacro Cuore, Policlinico Gemelli, unità operativa di Pneumologia, Roma, RM
  - Università Roma La Sapienza, servizio di Fisiopatologia respiratoria, Roma, RM
  - Università di Perugia -Terni, Medcina del lavoro Terni, Terni, TI
  - Università degli studi di Torino, Dipartimento di scienze biomediche ed oncologia umana, Torino, TO
  - Ospedale di Cattinara, unità operativa di pneumologia, Trieste, TS
  - Ospedale di Bussolengo, Unità operativa di Pneumologia, Bussolengo, VR
  - azienda universitaria-ospedaliera istituti ospitalieri di Verona, unità operativa di Allergologia, Verona, VR
  - Servizio Pneumologico ASL Brindisi, Brindisi
  - Seconda Università degli stuidi di Napoli, unità Operativa di Pneumologia, Napoli
  - Università di Roma Tor Vergata, unità di malattie dell'apparato Respiratorio, Roma

REFERENCES:
- [Derived] Papi A, Marku B, Scichilone N, Maestrelli P, Paggiaro P, Saetta M, Nava S, Folletti I, Bertorelli G, Bertacco S, Contoli M, Plebani M, Barbaro MPF, Spanevello A, Aliani M, Pannacci M, Morelli P, Beghe B, Fabbri LM; AIFASMA Study Group. Regular versus as-needed budesonide and formoterol combination treatment for moderate asthma: a non-inferiority, randomised, double-blind clinical trial. Lancet Respir Med. 2015 Feb;3(2):109-119. doi: 10.1016/S2213-2600(14)70266-8. Epub 2014 Dec 4. PMID 25481378